CLINICAL TRIAL: NCT03035955
Title: The Effect of Azelaic Acid (Financea Gel 15%) on Demodex Folliculorum Counts in Adult Subjects With Mild to Moderate Papulopustular Rosacea
Brief Title: Azelaic Acid on Demodex Counts in Rosacea
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00014511
Record Dates: First submitted 2012-12-19; First posted 2017-01-30 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-08

CONDITIONS: Rosacea
Keywords: Rosacea; Wake Forest; Demodex; Finacea Gel
MeSH Terms: conditions — Rosacea | interventions — azelaic acid

STUDY DESIGN:
Intervention Model Description: This is a split face, randomized, single blind, single center study. Male and female (non-pregnant, non-nursing) subjects, age 18 or greater, with mild to moderate papulopustular (based on Investigator Global Assessment) facial rosacea, with bilateral facial involvement, and no more than two nodules will be enrolled. Subjects will be randomized 1:1 by the study coordinator using a standard randomization table to receive azelaic acid (Finacea® Gel, 15%) twice daily on either the left side or the right side of the face and no treatment on the other side of the face.
Who Masked: Investigator
Masking Description: The investigator is blinded to which side of face is using the azelaeic acid treatetment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Azelaic acid (Active Comparator): azelaic acid (Finacea® Gel, 15%) twice daily on either the left side or the right side of the face and no treatment on the other side of the face
  Interventions: Drug: Azelaic acid
- no treatment (No Intervention): no treatment on the other side of the face

INTERVENTIONS:
Drug: Azelaic acid — 15% gel twice daily for four weeks to one side of face
  Other Names: Finacea Gel
  Arms: Azelaic acid

SUMMARY:
The purpose of this study is to measure the effects of azelaic acid on Demodex folliculorum counts and disease condition via a split face design in approximately twenty patients with mild to moderate rosacea. The investigators hypothesize that treatment of rosacea with azelaic acid will lead to a decreased Demodex folliculorum count as well as an improvement in lesion count and redness.

DETAILED DESCRIPTION:
This is a split face, randomized, single blind, single center study. Male and female (non-pregnant, non-nursing) subjects, age 18 or greater, with mild to moderate papulopustular facial rosacea, with bilateral facial involvement, and no more than two nodules will be enrolled. Subjects will be randomized 1:1 by the study coordinator using a standard randomization table to receive azelaic acid twice daily on either the left side or the right side of the face and no treatment on the other side of the face. Subjects must have a positive Demodex folliculorum standardized skin surface biopsy, defined at >5 mites cm at Screening/Baseline on at least one of two different SSSB specimens on bilateral sides of the face. The SSSB test location will ideally be on the cheek, but may be done in the most disease involved area. Subjects will be seen at Screening/Baseline, Week 1 and Week 4. Standard topical washout periods will be observed. At each visit, rosacea will be evaluated by lesion count, IGA and two Demodex SSSB tests done on each side of the face. Safety will be monitored at each visit using the Investigator Skin Irritation Assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, ages 18 and over, with mild to moderate paulopustular rosacea with bilateral facila involvement, who agrees to participate and provide written consent.
* Positive Demodex folliculorum SSSB, defined as >5 mites/cm on at least on of two different SSSB specimens on bilateral sides of teh face.
* Have an IGA of mild to moderate rosacea, rating between 2 and 5.

Exclusion Criteria:

* Use of topical therapy for rosacea or other skin conditions on the face within two weeks of Baseline.
* Use of oral medications for the treatment of rosacea that have been started or altered within the past three months.
* Presence of a concurrent medical condition or skin condition, which is determined by the investigator to potentially interfere with study outcomes or patient assessments.
* Subjects with known allergy or sensitivity to azelaic acid gel or components therein, such as propylene glycol.
* Subjects with known allergy or sensitivity to cyanoacrylates or formaldehyde.
* Presence of more than two nodules.
* Female subjects who are not postmenopausal for at least 1 year, surgically sterile or willing to practice effective contraception during the study. Reliable methods of birth control are: abstinence, oral contraceptives, intrauterine device, DepoProvera, tubal ligation or vasectomy of the partner in a monogamous relationship. An acceptable, though less reliable, method involves the careful use of condoms and spermicidal foam or gel and/or a cervical cap or sponge. Nursing mothers, pregnant women and women planning to become pregnant while on study are to be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02-02 (Actual); Study Completion 2012-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Fleischer, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Department of Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Azelaic Acid Left/No Treatment Right: azelaic acid (Finacea® Gel, 15%) twice daily on the left side side of the face and no treatment on the right side of the face
  Azelaic acid: 15% gel twice daily for four weeks to the left side of face
- Azelaic Acid Right/No Treatment Left: azelaic acid (Finacea® Gel, 15%) twice daily on the right side side of the face and no treatment on the left side of the face
  Azelaic acid: 15% gel twice daily for four weeks to the right side of face
Period: Overall Study
Arm/Group | Azelaic Acid Left/No Treatment Right | Azelaic Acid Right/No Treatment Left
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Azelaic Acid Left/No Treatment Right: azelaic acid (Finacea® Gel, 15%) twice daily on the left side side of the face and no treatment on the right side of the face
- Azelaic Acid Right/No Treatment Left: azelaic acid (Finacea® Gel, 15%) twice daily on the right side side of the face and no treatment on the left side of the face
- Total: Total of all reporting groups
Arm/Group | Azelaic Acid Left/No Treatment Right | Azelaic Acid Right/No Treatment Left | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Demodex Count
Description: number of demodex at Baseline and Week 4. Only Week 4 reported
Time Frame: Week 4
Measure: Number; unit: number of demodex
Groups:
- Azelaic Acid Right /no Treatment Left: azelaic acid (Finacea® Gel, 15%) twice daily on the right side side of the face and no treatment on the left side of the face
Arm/Group | Azelaic Acid Left/no Treatment Right | Azelaic Acid Right /no Treatment Left
Number analyzed (Participants) | 10 | 10
number of demodex | 40 | 18

ADVERSE EVENTS:
Arm/Group | Azelaic Acid | no Treatment
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes